CLINICAL TRIAL: NCT04992442
Title: A Phase 1 Study to Assess Absolute Bioavailability of TAK-935 (OV935) and to Characterize Mass Balance, Pharmacokinetics, Metabolism, and Excretion of [14C]TAK-935 (OV935) in Healthy Adult Male Participants
Brief Title: Study to Assess Absolute Bioavailability of TAK-935 (OV935) and to Characterize Mass Balance, Pharmacokinetics, Metabolism, and Excretion of [14C]TAK-935 (OV935) in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TAK-935-1008
Record Dates: First submitted 2021-08-03; First posted 2021-08-05 (Actual); Results first posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — soticlestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAK-935 300 mg + [14C]TAK-935 50 μg + [14C]TAK-935 300 mg (Experimental): TAK-935 3×100 mg, tablets, orally, once on Day 1, followed by [14C]TAK-935 50 micrograms (μg) [approximately 1 μCi], IV infusion, once on Day 1 of Treatment Period 1, followed by a Washout Period of 7 days, further followed by [14C]TAK-935 300 mg (approximately 100 μCi) solution, orally, once on Day 1 of Treatment Period 2.
  Interventions: Drug: TAK-935 Oral Tablet; Drug: [14C]TAK-935 IV Infusion; Drug: [14C]TAK-935 Oral Solution

INTERVENTIONS:
Drug: TAK-935 Oral Tablet — TAK-935 tablet
  Other Names: OV935; Soticlestat
Drug: [14C]TAK-935 IV Infusion — [14C]TAK-935 IV infusion
  Other Names: OV935
Drug: [14C]TAK-935 Oral Solution — [14C]TAK-935 oral solution
  Other Names: OV935

SUMMARY:
The purpose of this study is to determine absolute bioavailability (ABA) of TAK-935 (F) following a single microdose intravenous (IV) administration of 50 microgram (μg) (approximately 1 microcurie [μCi]) [14C]TAK-935 and a single oral administration of 3×100 mg milligram (mg) TAK-935 tablets in Treatment Period 1, and to assess the mass balance, characterize the pharmacokinetics (PK) of TAK-935 and metabolite [M-I (N-oxide)] in plasma and urine, and total radioactivity concentration equivalents in plasma and whole blood following a single oral administration of 300 mg (approximately 100 μCi) [14C]TAK-935 in Treatment Period 2.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-935 (also known as soticlestat/OV935). The study determines ABA in Treatment Period 1, and the absorption, metabolism, excretion, and mass balance of TAK-935 after single oral administration in Treatment Period 2 in healthy adult male participants, by collecting plasma, urine, and feces samples for drug concentration analysis, and plasma, whole blood, urine, and fecal samples for total radioactivity analysis and metabolic profiling.

The study will enroll approximately 6 healthy adult male participants. The study is designed to consist of 2 periods: Treatment Period 1 (ABA Study Period) and Treatment Period 2 (Absorption, Distribution, Metabolism, and Elimination [ADME] Study Period). In Treatment Period 1, all participants will receive a single unlabelled oral dose of TAK-935 as 3×100 mg tablets and a microdose IV infusion of 50 μg (approximately 1 μCi) [14C]TAK-935, followed by a Washout Period of 7 days before the dose in Treatment Period 2. In Treatment Period 2, all participants will receive a single dose of 300 mg (approximately 100 μCi) [14C]TAK-935 as an oral solution.

This single center trial will be conducted in the United States. The overall time to participate in this study is approximately 65 days including Screening Period. Participants will be contacted approximately 30 days after the last dose of study drug for a follow-up assessment. This compound was transferred to Takeda and acquired on 29 March 2021. This registration is retrospective due to the transfer of ownership.

ELIGIBILITY:
Inclusion Criteria:

1. Weighs at least 50 kg and body mass index (BMI) ≥18.0 and ˂32.0 kg/m^2 at Screening Visit.
2. Continuous nonsmoker who has not used nicotine-containing products (including vaping) for at least 3 months prior to the first dosing and throughout the study, based on participant self-reporting.
3. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the Investigator or designee.

Exclusion Criteria:

1. History or presence of cataracts or other clinically significant vision disturbances.
2. Abnormal and clinically significant ECG abnormality at Screening visit:

   * QT interval with Fridericia's correction method (QTcF) >450 milliseconds (ms) confirmed with one repeat testing.
3. History or presence of gastritis, gastrointestinal tract, gastric bypass surgery, or hepatic disorder or other clinical condition which, in the opinion of the Investigator or designee, may affect the absorption, distribution, metabolism, or elimination of study drug.
4. Has a risk of suicide according to the Investigator's clinical judgment [e.g., per Columbia-Suicide Severity Rating Scale (C-SSRS)] or has made a suicide attempt in the previous year prior to Screening Visit.
5. Positive urine drug or alcohol results at screening or first check-in.
6. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) or novel coronavirus 2019 (COVID-19).
7. Seated blood pressure is less than 90/40 millimeter of mercury (mmHg) or greater than 140/90 mmHg at Screening.
8. Seated HR is lower than 40 beats per minute (bpm) or higher than 99 bpm at Screening Visit.
9. Estimated creatinine clearance <80 mL/min at Screening Visit.
10. Has tattoo(s) or scarring at or near the site of IV infusion or any other condition which may interfere with infusion site examination, in the opinion of the Investigator.
11. Has infrequent bowel movements (less than approximately once per day) within 30 days prior to first dosing.
12. Recent history of abnormal bowel movements, such as diarrhea, loose stools, or constipation, within 2 weeks prior to first dosing.
13. Has received radiolabeled substances or has been exposed to radiation sources within 12 months of first dosing or is likely to receive radiation exposure or radioisotopes within 12 months of first dosing such that participation in this study would increase their total exposure beyond the recommended levels considered safe [i.e., weighted annual limit recommended by the International Commission on Radiological Protection (ICRP) of 3000 milli roentgen equivalent man (mrem)].
14. Unable to refrain from or anticipates the use of:

    1. Any drug, including prescription and nonprescription medications, herbal remedies, or vitamin supplements within 14 days prior to the first dosing and throughout the study, including the Follow-up Period. Thyroid hormone replacement medication may be permitted if the participant has been on the same stable dose for the immediate 3 months prior to first study drug administration. After the first dose of study drug, ibuprofen (up to 1.2 g per 24 hours) may be administered at the discretion of the Investigator or designee. Milk of Magnesia (i.e., magnesium hydroxide) (≤60 mL per day) may be administered to ensure defecation, at discretion of the Investigator or designee.
    2. Any drugs known to be significant inducers of cytochrome P450 (CYP)3A4, CYP2C19 or uridine diphosphate glucuronosyltransferase (UGT), including St. John's Wort, within 28 days prior to the first dosing and throughout the study, including the Follow-up Period. Appropriate sources (e.g., Flockhart Table^TM) will be consulted to confirm lack of PK/pharmacodynamic interaction with study drug(s).
    3. Alcohol
15. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
16. Donation of blood or significant blood loss within 56 days prior to the first dosing.
17. Plasma donation within 7 days prior to the first dosing.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 09 July 2020 to 18 August 2020.
Pre-assignment Details: Healthy male participants were enrolled in this study to receive TAK-935 tablets followed by radio-labelled TAK-935 intravenous (IV) infusion on Day 1 of Treatment Period 1 and radio-labelled TAK-935 oral solution on Day 1 of Treatment Period 2. There was a 7-day Washout Period between the two periods.
Period: Treatment Period 1
Arm/Group | TAK-935 300 mg + [14C]TAK-935 50 μg + [14C]TAK-935 300 mg
Started | 6
Completed | 6
Not Completed | 0
Period: Washout Period
Arm/Group | TAK-935 300 mg + [14C]TAK-935 50 μg + [14C]TAK-935 300 mg
Started | 6
Completed | 6
Not Completed | 0
Period: Treatment Period 2
Arm/Group | TAK-935 300 mg + [14C]TAK-935 50 μg + [14C]TAK-935 300 mg
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least one dose of the study drug.
Groups:
- TAK-935 300 mg + [14C]TAK-935 50 μg + [14C]TAK-935 300 mg: TAK-935 3×100 mg, tablets, orally, once on Day 1, followed by [14C]TAK-935 50 μg [approximately 1 μCi], IV infusion, once on Day 1 of Treatment Period 1, followed by a Washout Period of 7 days, further followed by [14C]TAK-935 300 mg (approximately 100 μCi) solution, orally, once on Day 1 of Treatment Period 2.
Arm/Group | TAK-935 300 mg + [14C]TAK-935 50 μg + [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (14.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6
Weight [Mean (Standard Deviation); unit: kg] | 84.82 (16.899)
Height [Mean (Standard Deviation); unit: cm] | 176.5 (7.31)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI = Weight (kg)/Height (m)^2
  kg/m^2 | 27.000 (3.4142)

OUTCOME MEASURES:

1. Primary Outcome: Period 1: Percent Absolute Bioavailability (%F) for TAK-935
Description: Bioavailability is defined as the proportion of a drug which enters the circulation when introduced into the body and so is able to have an active effect. Percent absolute bioavailability, calculated for plasma TAK-935 as [Actual Dose (IV) x Area Under the Concentration-time Curve from Time 0 to Infinity {AUCinf} (oral)] / [Actual Dose (oral) x AUCinf (IV)] x 100.
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose in Treatment Period 1
Population: Pharmacokinetic (PK) Population included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received the oral dose of TAK-935 3×100 mg tablets and 50 μg IV dose in Treatment Period 1 were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent absolute bioavailability
Groups:
- TAK-935 300 mg + [14C]TAK-935 50 μg: TAK-935 3×100 mg tablets, orally, followed by [14C]TAK-935 50 μg (approximately 1 μCi), 15-minute IV infusion, once on Day 1 of Treatment Period 1.
Arm/Group | TAK-935 300 mg + [14C]TAK-935 50 μg
Number analyzed (Participants) | 6
percent absolute bioavailability | 12.57 (75.1)

2. Primary Outcome: Period 2: Total Radioactivity Expressed as Cumulative Percentage of Dose of [14C]TAK-935 Excreted in Urine and Feces Combined [Combined Cum%Dose]
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: PK Population included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received the dose of [14C]TAK-935 300 mg oral solution in Treatment Period 2 were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Groups:
- [14C]TAK-935 300 mg: [14C]TAK-935 300 mg (approximately 100 μCi), solution, orally, under fasted state, once on Day 1 of Treatment Period 2.
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
percentage of dose | 97.55 (0.5)

3. Primary Outcome: Period 2: Total Radioactivity Expressed as Amount of [14C]TAK-935 Excreted in Urine (CumAe[u])
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: Analysis Population Description: PK Population included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received the dose of [14C]TAK-935 300 mg oral solution in Treatment Period 2 were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg equivalents (eq) of parent drug
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
mg equivalents (eq) of parent drug | 292.3 (1.4)

4. Primary Outcome: Period 2: Total Radioactivity Expressed as Amount of [14C]TAK-935 Excreted in Feces (CumAe[f])
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg eq of parent drug
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
mg eq of parent drug | 9.429 (48.2)

5. Primary Outcome: Period 2: Total Radioactivity Expressed as Amount of [14C]TAK-935 Excreted in Urine and Feces Combined (Combined CumAe)
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg eq of parent drug
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
mg eq of parent drug | 300.7 (0.5)

6. Primary Outcome: Period 2: Percentage of Administered Radioactive Dose of [14C]TAK-935 Excreted in Urine (Cum%Dose[u])
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
percentage of dose | 94.81 (1.4)

7. Primary Outcome: Period 2: Percentage of Administered Radioactive Dose of [14C]TAK-935 Excreted in Feces (Cum%Dose[f])
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
percentage of dose | 3.058 (48.2)

8. Primary Outcome: Period 2: Cmax: Maximum Observed Plasma Concentration of TAK-935
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
ng/mL | 1352 (61.3)

9. Primary Outcome: Period 2: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) of TAK-935
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
hours (hr) | 0.42 [0.42 to 0.42]

10. Primary Outcome: Period 2: t(1/2)z: Terminal Disposition Phase Half-life of TAK-935 in Plasma
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: PK Population included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received the dose of [14C]TAK-935 300 mg oral solution in Treatment Period 2 were evaluated for this outcome measure. Overall number analyzed is the number of participants with data available for analysis.
Measure: Median (Full Range); unit: hr
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 5
hr | 4.374 [3.51 to 10.55]

11. Primary Outcome: Period 2: AUC0-inf: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity of TAK-935
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 5
ng*hr/mL | 1805 (40.4)

12. Primary Outcome: Period 2: AUC0-t: Area Under the Plasma Concentration-time Curve From Time 0 to Time t for TAK-935
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
ng*hr/mL | 1547 (40.8)

13. Primary Outcome: Period 2: AUC0-last: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration of TAK-935
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
ng*hr/mL | 1638 (43.1)

14. Primary Outcome: Period 2: Cmax: Maximum Observed Plasma Radioactivity Concentration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq/mL
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
ng eq/mL | 17220 (34.4)

15. Primary Outcome: Period 2: Tmax: Time to Reach the Maximum Plasma Radioactivity Concentration (Cmax)
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hr
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
hr | 0.599 [0.43 to 0.77]

16. Primary Outcome: Period 2: t(1/2)z: Terminal Disposition Phase Half-life of Plasma Radioactivity Concentration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
hr | 3.655 [2.78 to 10.82]

17. Primary Outcome: Period 2: AUC0-inf: Area Under the Plasma Radioactivity Concentration-time Curve From Time 0 to Infinity
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq*hr/mL
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
ng eq*hr/mL | 42890 (21.4)

18. Primary Outcome: Period 2: AUC0-t: Area Under the Plasma Radioactivity Concentration-time Curve From Time 0 to Time t
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq*hr/mL
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
ng eq*hr/mL | 39580 (21.6)

19. Primary Outcome: Period 2: AUC0-last: Area Under the Plasma Radioactivity Concentration-time Curve From Time 0 to Last Quantifiable Concentration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq*hr/mL
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
ng eq*hr/mL | 40650 (21.9)

20. Primary Outcome: Period 2: Cmax: Maximum Observed Whole Blood Radioactivity Concentration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq/g
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
ng eq/g | 9157 (29.0)

21. Primary Outcome: Period 2: Tmax: Time to Reach the Maximum Whole Blood Radioactivity Concentration (Cmax)
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
hr | 0.440 [0.44 to 0.77]

22. Primary Outcome: Period 2: t(1/2)z: Terminal Disposition Phase Half-life of Whole Blood Radioactivity Concentration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
hr | 3.678 [3.04 to 20.42]

23. Primary Outcome: Period 2: AUC0-inf: Area Under the Whole Blood Radioactivity Concentration-time Curve From Time 0 to Infinity
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms (ng) eq*hr/g
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
nanograms (ng) eq*hr/g | 24420 (19.9)

24. Primary Outcome: Period 2: AUC0-t: Area Under the Whole Blood Radioactivity Concentration-time Curve From Time 0 to t
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: The data for TAK-935 concentration in whole blood were not collected therefore AUC0-t cannot be determined and not available.
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 0

25. Primary Outcome: Period 2: AUC0-last: Area Under the Whole Blood Radioactivity Concentration-time Curve From Time 0 to Last Quantifiable Concentration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq*hr/g
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
ng eq*hr/g | 22280 (20.2)

26. Primary Outcome: Period 2: CLR: Renal Clearance for TAK-935 in Urine
Description: Renal clearance (CLr) is the volume of plasma entering the kidney that is completely cleared of drug per unit of time.
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
L/hr | 6.792 (21.8)

27. Primary Outcome: Period 2: Aet1-t2: Amount of TAK-935 Excreted in the Urine in Each Collection Interval
Time Frame: 0-12, 12-24, 24-48, 48-72, 72-96, 96-120 hours post-dose in Treatment Period 2
Population: PK Population included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received the dose of [14C]TAK-935 300 mg oral solution in Treatment Period 2, with data available for analysis at the given timepoint were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg eq
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
mg eq
  Ae0-12 hours | 268.1 (4.4)
  Ae12-24 hours | 18.28 (35.0)
  Ae24-48 hours | 3.829 (66.2)
  Ae48-72 hours | 0.3126 (92.8)
  Ae72-96 hours | 0.1946 (80.6)
  Ae96-120 hours: number analyzed (Participants) | 1
  Ae96-120 hours | 0.2296 (NA) — The geometric coefficient of variation was not estimable as only one participant had measurable amount.

28. Primary Outcome: Period 2: Whole Blood to Plasma Partitioning Ratio: Change From Baseline in Percentage of [14C]TAK-935 Radioactivity in Whole Blood Relative to Plasma
Time Frame: 0.17, 0.42, 0.75, 1.5, 2.5, 4.5, 8, 12, and 24 hours post-dose in Treatment Period 2
Population: PK Population included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received the dose of [14C]TAK-935 300 mg oral solution in Treatment Period 2 were evaluated for this outcome measure. Number analyzed are the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6
ratio
  0.17 Hour | 0.5881 (0.065712)
  0.42 Hour | 0.5440 (0.054836)
  0.75 Hour | 0.5561 (0.026316)
  1.5 Hours | 0.5361 (0.025054)
  2.5 Hours | 0.5934 (0.052200)
  4.5 Hours | 0.5823 (0.038252)
  8 Hours | 0.5647 (0.046592)
  12 Hours | 0.6960 (0.16172)
  24 Hours: number analyzed (Participants) | 1
  24 Hours | 1.036 (NA) — The standard deviation was not estimable as there was only one participant.

29. Secondary Outcome: Period 1: Ceoi: Plasma Concentration at the End of Infusion for [14C]TAK-935
Time Frame: Day 1: At the end of infusion (at 15 minutes post dose) in Treatment Period 1
Population: PK Population included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received [14C]TAK-935 50 μg IV infusion in Treatment Period 1 were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms (pg) eq /mL
Groups:
- [14C]TAK-935 50 μg: [14C]TAK-935 50 μg (approximately 1 μCi), infusion, 15-minute IV infusion, once on Day 1 of Treatment Period 1 after the TAK-935 oral dose, followed by a Washout Period of at least 7 days.
Arm/Group | [14C]TAK-935 50 μg
Number analyzed (Participants) | 6
picograms (pg) eq /mL | 2472 (22.7)

30. Secondary Outcome: Period 1: Cmax: Maximum Observed Plasma Concentration for TAK-935 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose in Treatment Period 1
Population: PK Population included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received the oral dose of TAK-935 3×100 mg tablets in Treatment Period 1 were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- TAK-935 300 mg: TAK-935 3×100 mg tablets, orally, once on Day 1 of Treatment Period 1.
Arm/Group | TAK-935 300 mg
Number analyzed (Participants) | 6
ng/mL | 822.8 (149.6)

31. Secondary Outcome: Period 1: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-935 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose in Treatment Period 1
Population: as for outcome 30
Measure: Median (Full Range); unit: hr
Arm/Group | TAK-935 300 mg
Number analyzed (Participants) | 6
hr | 1.129 [0.42 to 1.54]

32. Secondary Outcome: Period 1: AUC0-inf: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-935 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose in Treatment Period 1
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | TAK-935 300 mg
Number analyzed (Participants) | 6
ng*hr/mL | 1304 (69.3)

33. Secondary Outcome: Period 1: AUC0-inf: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for [14C]TAK-935 After IV Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 47.5 hours) post-dose in Treatment Period 1
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg eq*hr/mL
Arm/Group | [14C]TAK-935 50 μg
Number analyzed (Participants) | 6
pg eq*hr/mL | 1742 (15.1)

34. Secondary Outcome: Period 1: AUC0-t: Area Under the Plasma Concentration-time Curve From Time 0 to t After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose in Treatment Period 1
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | TAK-935 300 mg
Number analyzed (Participants) | 6
ng*hr/mL | 1250 (68.6)

35. Secondary Outcome: Period 1: AUC0-t: Area Under the Plasma Concentration-time Curve From Time 0 to Time t for TAK-935 After IV Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 47.5 hours) post-dose in Treatment Period 1
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg eq*hr/mL
Arm/Group | [14C]TAK-935 50 μg
Number analyzed (Participants) | 6
pg eq*hr/mL | 1691 (15.1)

36. Secondary Outcome: Period 1: AUC0-last: Area Under the Plasma Concentration-time Curve From Time 0 to Last Quantifiable Concentration for TAK-935 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose in Treatment Period 1
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | TAK-935 300 mg
Number analyzed (Participants) | 6
ng*hr/mL | 1268 (70.3)

37. Secondary Outcome: Period 1: AUC0-last: Area Under the Plasma Concentration-time Curve From Time 0 to Last Quantifiable Concentration for [14C]TAK-935 After IV Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 47.5 hours) post-dose in Treatment Period 1
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg eq*hr/mL
Arm/Group | [14C]TAK-935 50 μg
Number analyzed (Participants) | 6
pg eq*hr/mL | 1713 (15.3)

38. Secondary Outcome: Period 1: t(1/2)z: Terminal Disposition Half-life for TAK-935 After Oral Administration in Plasma
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 30
Measure: Median (Full Range); unit: hr
Arm/Group | TAK-935 300 mg
Number analyzed (Participants) | 6
hr | 4.249 [2.19 to 5.95]

39. Secondary Outcome: Period 1: t(1/2)z: Terminal Disposition Half-life for [14C]TAK-935 After IV Administration in Plasma
Time Frame: Day 1 pre-dose and at multiple time points (up to 47.5 hours) post-dose
Population: as for outcome 29
Measure: Median (Full Range); unit: hr
Arm/Group | [14C]TAK-935 50 μg
Number analyzed (Participants) | 6
hr | 1.358 [0.60 to 12.46]

40. Secondary Outcome: Period 1: Total Radioactivity Expressed as Amount of [14C]TAK-935 Excreted in Urine (CumAe[u]) After IV Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 1
Population: PK Population included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received [14C]TAK-935 50 μg IV infusion in Treatment Period 1 were evaluated for this outcome measure. Overall number analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg eq
Arm/Group | [14C]TAK-935 50 μg
Number analyzed (Participants) | 5
µg eq | 48.14 (1.4)

41. Secondary Outcome: Period 1: Total Radioactivity Expressed as Amount of [14C]TAK-935 Excreted in Feces (CumAe[f]) After IV Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 1
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg eq
Arm/Group | [14C]TAK-935 50 μg
Number analyzed (Participants) | 6
µg eq | 0.7988 (76.2)

42. Secondary Outcome: Period 1: Total Radioactivity Expressed as Amount of [14C]TAK-935 Excreted in Urine and Feces Combined (Combined CumAe) After IV Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 1
Population: as for outcome 40
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg eq
Arm/Group | [14C]TAK-935 50 μg
Number analyzed (Participants) | 5
µg eq | 48.82 (1.4)

43. Secondary Outcome: Period 1: Percentage of Administered Radioactive Dose of [14C]TAK-935 Excreted in Urine (Cum%Dose[u]) After IV Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 1
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | [14C]TAK-935 50 μg
Number analyzed (Participants) | 6
percentage of dose | 95.17 (1.3)

44. Secondary Outcome: Period 1: Percentage of Administered Radioactive Dose of [14C]TAK-935 Excreted in Feces (%Dose[f]) After IV Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 1
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | [14C]TAK-935 50 μg
Number analyzed (Participants) | 6
percentage of dose | 1.587 (76.4)

45. Secondary Outcome: Period 2: Metabolic Profile of TAK-935 in Plasma After Oral Administration of [14C]TAK-935
Description: The metabolic profile of TAK-935 after oral administration of [14C]TAK-935 was done to assess the presence of TAK-935 and various metabolites (M1 to M9) in plasma in at least one sample using radiometric detection and/or liquid chromatography mass spectroscopy (LCMS). The presence of any metabolite is indicated as '1' and absence is indicated as '0'. Only categories with value '1' are reported.
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Number; unit: sample positive
Groups:
- [14C]TAK-935 300 mg (Plasma): [14C]TAK-935 300 mg (approximately 100 μCi), solution, orally, under fasted state, once on Day 1 of Treatment Period 2.
Arm/Group | [14C]TAK-935 300 mg (Plasma)
Number analyzed (Participants) | 6
sample positive
  TAK-935 | 1
  M1 | 1
  M2 | 0
  M3 | 1
  M4 | 1
  M5 | 0
  M6 | 0
  M7 | 0
  M8 | 1
  M9 | 0

46. Secondary Outcome: Period 2: Metabolic Profile of TAK-935 in Urine and Feces After Oral Administration of [14C]TAK-935
Description: The metabolic profile of TAK-935 after oral administration of [14C]TAK-935 was done to assess the presence of TAK-935 and various metabolites (M1 to M9) in urine and feces in at least one sample using radiometric detection and/or LCMS. The presence of any metabolite is indicated as '1' and absence is indicated as '0'. Data is reported separately for urine and feces.
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Number; unit: sample positive
Groups:
- [14C]TAK-935 300 mg (Urine); [14C]TAK-935 300 mg (Feces): [14C]TAK-935 300 mg (approximately 100 μCi), solution, orally, under fasted state, once on Day 1 of Treatment Period 2.
Arm/Group | [14C]TAK-935 300 mg (Urine) | [14C]TAK-935 300 mg (Feces)
Number analyzed (Participants) | 6 | 6
sample positive
  TAK-935 | 1 | 1
  M1 | 1 | 0
  M2 | 1 | 1
  M3 | 1 | 0
  M4 | 1 | 0
  M5 | 1 | 0
  M6 | 1 | 0
  M7 | 1 | 0
  M8 | 1 | 1
  M9 | 0 | 1

47. Secondary Outcome: Percentage of Participants Reporting One or More Treatment Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an AE that is starting or worsening at the time of or after study drug administration.
Time Frame: From first dose up to 30 days after last dose of study drug (up to approximately 40 days)
Population: Safety Population included all participants who received at least one dose of the study drug. As prespecified in the protocol data for adverse events was collected and reported for Period 1 and Period 2.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-935 300 mg + [14C]TAK-935 50 μg | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6 | 6
percentage of participants | 0 | 16.7

48. Secondary Outcome: Percentage of Participants With Treatment Emergent Clinically Relevant Changes in Electrocardiogram (ECG) Parameters
Time Frame: From first dose up to 30 days after last dose of study drug (up to approximately 40 days)
Population: Safety Population included all participants who received at least one dose of the study drug. As prespecified in the protocol data for this outcome measure was collected and reported for Period 1 and Period 2.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-935 300 mg + [14C]TAK-935 50 μg | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6 | 6
percentage of participants | 0 | 0

49. Secondary Outcome: Percentage of Participants With Treatment Emergent Clinically Relevant Changes in Vital Sign Parameters
Description: Vital Signs included blood pressure (systolic and diastolic), heart rate (HR), respiratory rate, and temperature.
Time Frame: From first dose up to 30 days after last dose of study drug (up to approximately 40 days)
Population: as for outcome 48
Measure: Number; unit: percentage of participants
Arm/Group | TAK-935 300 mg + [14C]TAK-935 50 μg | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6 | 6
percentage of participants | 0 | 0

50. Secondary Outcome: Percentage of Participants With Treatment Emergent Clinically Relevant Changes in Laboratory Parameters
Description: The laboratory parameters included tests for serum chemistry, hematology, coagulation, and urinalysis.
Time Frame: From first dose up to 30 days after last dose of study drug (up to approximately 40 days)
Population: as for outcome 48
Measure: Number; unit: percentage of participants
Arm/Group | TAK-935 300 mg + [14C]TAK-935 50 μg | [14C]TAK-935 300 mg
Number analyzed (Participants) | 6 | 6
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose up to 30±2 days after last dose of study drug (up to approximately 40 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory/exam findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety Population included all participants who received at least one dose of the study drug. As prespecified in the protocol data for adverse events was collected and reported for Period 1 and Period 2.
Arm/Group | TAK-935 300 mg + [14C]TAK-935 50 μg | [14C]TAK-935 300 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-935 300 mg + [14C]TAK-935 50 μg (N=6) | [14C]TAK-935 300 mg (N=6)
Headache (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT04992442/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT04992442/SAP_001.pdf